CLINICAL TRIAL: NCT05404061
Title: Why do Some Patients Respond Better Than Others to Bariatric Surgery?
Brief Title: The Poor Responders Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Imperial College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 17/LO/1323
Record Dates: First submitted 2022-03-08; First posted 2022-06-03 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Bariatric Surgery Candidate; Obesity, Morbid; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Obesity, Morbid; Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gut hormone secretion study (No Intervention): This will be a retrospective study of participants who have undergone bariatric surgery. On the day of the visit participants will undergo comprehensive physiological profiling which will include the following tests:
  * Body weight and bioelectrical impedance analysis
  * Mixed Meal Tolerance Test. This will be analysed for metabolites including gut hormones, insulin, glucose, bile acids and their sub-fractions, fibroblast-growth factors, lipids and immune profiles.
  * Resting Energy Expenditure and Diet Induced Thermogenesis assessed via Indirect Calorimetry
  * Metabolomic and Metagenomic Assessment
- Gut hormone sensitivity study (Placebo Comparator): This will be a single blinded study with participants attending three visits. Their first visit will act as an acclimatisation visit and participants will be infused subcutaneously with a triple gut hormone infusion (GLP-1, PYY and OXM). This will not only allow us to acclimatise the study volunteer to the study visits, but also allow us to test for subject tolerability of the gut hormones. Occasionally some volunteers are more sensitive to the gut hormone infusion and the doses needs to be titrated down. The doses used will be established doses of the gut hormones infused previously and which have been shown to be safe and tolerated, and to reduce appetite (In house data).
  Interventions: Other: Gut hormones
- Prospective assessment of gut hormone response pre and post-surgery (No Intervention): This will be a prospective study assessing the gut hormone response pre and post bariatric surgery.
  On the day of the visit participants will undergo comprehensive physiological profiling which will include the following tests:
  * Body weight and bioelectrical impedance analysis
  * Mixed Meal Tolerance Test. This will be analysed for metabolites including gut hormones, insulin, glucose, bile acids and their sub-fractions, fibroblast-growth factors, lipids and immune profiles.
  * Resting Energy Expenditure and Diet Induced Thermogenesis assessed via Indirect Calorimetry
  * Metabolomic and Metagenomic Assessment

INTERVENTIONS:
Other: Gut hormones — Their first visit will act as an acclimatisation visit and participants will be infused subcutaneously with a triple gut hormone infusion (GLP-1, PYY and OXM). This will not only allow us to acclimatise the study volunteer to the study visits, but also allow us to test for subject tolerability of the gut hormones.
  For the next two visits participants will be randomised in a single-blinded fashion to a subcutaneous infusion of either:
  1. 0.9% saline,
  2. GLP-1
  Arms: Gut hormone sensitivity study

SUMMARY:
Obesity and type 2 diabetes are major causes of illness and premature death worldwide and their incidence is increasing rapidly. Bariatric surgery is considered as the "gold-standard" surgical treatment for both conditions.

However, not all patients do equally well after surgery and indeed the weight loss experienced by patients undergoing bariatric surgery can vary. As such when patients are seen after bariatric surgery in clinic they fall in one of the following two categories:

1. Good responders: this is the majority of patients who lose the expected amount of weight based on the published studies.
2. Poor responders: this is a small group of patients who either lose less than the expected amount of weight after bariatric surgery or lose the expected amounts of weight early after surgery but then regain a substantial proportion of the weight they have lost.

The so-called "poor responders" are exposed to all the risks of the operation and do not benefit from the weight loss as much as good responders.

This study would therefore like to investigate the physiological factors that distinguish poor from good responders before, and after bariatric surgery. The study team hypothesizes that compared to good responders, poor responders exhibit:

1. a smaller degree of fullness sensation after a meal,
2. a lower energy expenditure after a meal, and
3. genetic changes (single nucleotide polymorphisms) that predispose the poor responder to development of obesity.

In addition, the study team hypothesizes that poor responders exhibit:

1. lower gut hormone secretion after a meal and
2. are less sensitive to the physiological action of gut hormones compared to good responders and that this difference in gut hormone secretion and response to gut hormones prior to bariatric surgery can be helpful to predict response to bariatric surgery.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 -70 years.
* Male or female.
* Previous bariatric surgery for obesity and/or diabetes (studies 1 and 2).
* ≥1 year interval after bariatric surgery (studies 1 and 2).
* Awaiting bariatric surgery at the Imperial Weight Centre (study 3)
* Able to give informed consent.

Exclusion Criteria:

* History of any medical, psychological or other condition, or use of any medications, including over-the-counter products, which, in the opinion of the investigators, would either interfere with the study or potentially cause harm to the volunteer.
* Without access at home to a telephone or other factor likely to interfere with ability to participate reliably in the study.
* Pregnancy or breastfeeding.
* Unable to maintain adequate contraception for the duration of the study and for one month afterwards.
* History of hypersensitivity to any of the components of the subcutaneous infusions.
* Donated blood during the preceding 3 months or intention to do so before the end of the study.
* Any other co-morbidity that would compromise the validity of the study or the safety of the participant such as heart failure or clinically apparent cardiovascular disease.
* Anatomical or endocrinological pathology causing poor weight loss or weight regain
* Uncontrolled hypertension (systolic blood pressure of 160 mmHg or above and/or diastolic blood pressure of 100 mmHg or above)
* Participation in a research study within the last two months.
* Unable to speak English (this is relevant to answering the psychological questionnaires)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2027-09-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Gut hormone secretion study: Peak plasma level of gut hormones after meal ingestion | During one study visit (Mixed Meal Test), at least 1 year post-surgery.
  A standardized mixed-meal tolerance test. Blood samples will be taken at intervals over four hours. These will be analysed for gut hormones.
Gut hormone sensitivity study: Change in Food intake following gut hormone infusion compared to placebo. | During three study visits (gut hormone infusion visits), at least 1 year post-surgery.
  Ad libitum meal test. A meal will be served to participants and they will be allowed 20 minutes to eat until they feel comfortably full. Food intake will be measured at the end of the meal.
Prospective assessment of gut hormone response pre and post-surgery: Change in Peak plasma level of gut hormones after meal ingestion. | During two study visits (Mixed Meal Test), one before and one 1 year after surgery.
  A standardized mixed-meal tolerance test. Blood samples will be taken at intervals over four hours. These will be analysed for gut hormones.

SECONDARY OUTCOMES:
Change in Resting Energy Expenditure | Change between two visits: before and 1 year after bariatric surgery (Prospective assessment of gut hormone response pre and post-surgery).
  Resting energy expenditure assessment via indirect calorimetry.
Change in Diet Induced Thermogenesis | Change between two visits: before and 1 year after bariatric surgery (Prospective assessment of gut hormone response pre and post-surgery).
  Diet induced thermogenesis assessment via indirect calorimetry.
Change in Genetic factors | Change between two visits: Before and 1 year after bariatric surgery.
  Change in genetic factors assessed by collection of plasma DNA samples.

CONTACTS AND LOCATIONS:
Overall Officials: Tricia M Tan, PhD, Principal Investigator — Imperial College London
Locations (1):
- Imperial College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aasheim ET, Aylwin SJ, Radhakrishnan ST, Sood AS, Jovanovic A, Olbers T, le Roux CW. Assessment of obesity beyond body mass index to determine benefit of treatment. Clin Obes. 2011 Apr;1(2-3):77-84. doi: 10.1111/j.1758-8111.2011.00017.x. Epub 2011 Jul 5. PMID 25585572
- [Background] Batterham RL, Cowley MA, Small CJ, Herzog H, Cohen MA, Dakin CL, Wren AM, Brynes AE, Low MJ, Ghatei MA, Cone RD, Bloom SR. Gut hormone PYY(3-36) physiologically inhibits food intake. Nature. 2002 Aug 8;418(6898):650-4. doi: 10.1038/nature00887. PMID 12167864
- [Background] De Silva A, Salem V, Long CJ, Makwana A, Newbould RD, Rabiner EA, Ghatei MA, Bloom SR, Matthews PM, Beaver JD, Dhillo WS. The gut hormones PYY 3-36 and GLP-1 7-36 amide reduce food intake and modulate brain activity in appetite centers in humans. Cell Metab. 2011 Nov 2;14(5):700-6. doi: 10.1016/j.cmet.2011.09.010. Epub 2011 Oct 13. PMID 22000927
- [Background] Laferrere B, Swerdlow N, Bawa B, Arias S, Bose M, Olivan B, Teixeira J, McGinty J, Rother KI. Rise of oxyntomodulin in response to oral glucose after gastric bypass surgery in patients with type 2 diabetes. J Clin Endocrinol Metab. 2010 Aug;95(8):4072-6. doi: 10.1210/jc.2009-2767. Epub 2010 May 25. PMID 20501690
- [Background] Tan TM, Field BC, McCullough KA, Troke RC, Chambers ES, Salem V, Gonzalez Maffe J, Baynes KC, De Silva A, Viardot A, Alsafi A, Frost GS, Ghatei MA, Bloom SR. Coadministration of glucagon-like peptide-1 during glucagon infusion in humans results in increased energy expenditure and amelioration of hyperglycemia. Diabetes. 2013 Apr;62(4):1131-8. doi: 10.2337/db12-0797. Epub 2012 Dec 17. PMID 23248172